CLINICAL TRIAL: NCT00550979
Title: Gestational Diabetes Mellitus and Implications for Cardiovascular Disease Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Rhonda Bentley-Lewis, MD, Rhonda Bentley-Lewis, MD, MBA, MMSc, Brigham and Women's Hospital
Other Study IDs: 2007P001406
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; cardiovascular disease risk; heart disease risk
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Black women with history of pregnancy/ies complicated by gestational diabetes mellitus
- 2: Black women with history of normal, uncomplicated pregnancy/ies
- 3: White women with a history of pregnancy/ies complicated by gestational diabetes.
- 4: White women with a history of normal, uncomplicated pregnancy/ies.

SUMMARY:
The purpose of this research study is to look at whether there are differences in blood vessel function, risk for developing diabetes (high blood sugar), lipid (blood fat) levels, and levels of other blood markers in women who have had a pregnancy complicated by diabetes as compared with women who have had a normal pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of self-identified African descent (black) and European (white) ancestry
* 18-40 years of age
* Regular menstrual cycles
* 5 or less years postpartum
* Have either a normal or a GDM index pregnancy history
* Are in good health free of thyroid, cardiac, or renal disease

Exclusion Criteria:

* If you are pregnant
* If you are lactating

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Black and white women who have had uncomplicated pregnancies or pregnancies complicated by gestational diabetes in the past 5 years
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2007-09; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
endothelial function | same day

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Bentley-Lewis, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts